CLINICAL TRIAL: NCT03157466
Title: Diaphragmatic Efficiency After Thyroid Hormone Replacement Therapy in Ventilated Patients With the Nonthyroidal Illness Syndrome: a Physiological Study
Brief Title: Respiratory Muscle Function After Thyroid Hormone Replacement Therapy in Nonthyroidal Illness Syndrome
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, BELLO GIUSEPPE, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 002
Record Dates: First submitted 2017-05-12; First posted 2017-05-17 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Thyroid Diseases; Respiratory Failure
MeSH Terms: conditions — Thyroid Diseases; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although it is now recognized that a variety of respiratory abnormalities, such as diaphragmatic dysfunction, can be present in primary hypothyroidism and reverse with adequate hormone treatment, the role of thyroid hormone replacement therapy on respiratory system in patients with the nonthyroidal illness syndrome (NTIS) remains to be clarified. The NTIS has been found to be an independent risk factor for prolonged (> 13 days) mechanical ventilation. It is unclear, however, whether the NTIS is only a biochemical prognostic marker or it actually contributes to the development and progression of respiratory failure.

The aim of this study will be to assess respiratory muscle function after thyroid hormone substitution therapy in mechanically ventilated patients with the NTIS.

ELIGIBILITY:
Inclusion Criteria:

* Patients under mechanical ventilation for more than 48 hours who experience a spontaneous breathing trial and have a diagnosis of nonthyroidal illness syndrome

Exclusion Criteria:

* • age <18 yr;

  * pregnancy or estro-progestinic therapy;
  * tracheostomy;
  * neurological or neuromuscular pathology and/or known phrenic nerve dysfunction;
  * previously diagnosed intrinsic thyroid disease; known or suspected pituitary-hypothalamic disease;
  * severe obesity;
  * ischemic cardiopathy; complex ventricular arrhythmias;
  * serum cortisol level below 80 ng/ml; renal or hepatic failure (respectively, creatininemia ≥ 3.5 mg/dL and bilirubinemia ≥ 6.0 mg/dL);
  * transfusion of plasma within 48 h prior to thyroid hormone assessment; use of amiodarone in the previous 8 weeks;
  * use of iodine contrast agents in the previous 8 weeks;
  * hemodialysis;
  * expected poor outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care unit and mechanically ventilated for more than 48 hours who fail weaining from ventilator and with a diagnosis of nonthyroidal illness syndrome
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline neuromechanical efficiency (obtained immediately before starting thyroid hormone therapy) at 3, 6, and 24 hours | 24 hours (study points at 3, 6, and 24 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, Italy

REFERENCES:
- [Derived] Bello G, Spinazzola G, Giammatteo V, Montini L, De Pascale G, Bisanti A, Annetta MG, Troiani E, Bianchi A, Pontecorvi A, Pennisi MA, Conti G, Antonelli M. Effects of Thyroid Hormone Treatment on Diaphragmatic Efficiency in Mechanically Ventilated Subjects With Nonthyroidal Illness Syndrome. Respir Care. 2019 Oct;64(10):1199-1207. doi: 10.4187/respcare.06770. Epub 2019 Apr 23. PMID 31015389